CLINICAL TRIAL: NCT04011345
Title: Folic Acid Supplementation in Children With Sickle-Cell Disease: A Randomized Double-Blind Cross-Over Trial
Brief Title: Folic Acid Supplementation in Children With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Crystal Karakochuk, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H18-02981
Record Dates: First submitted 2019-04-30; First posted 2019-07-08 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Anemia, Sickle Cell
Keywords: Folic Acid; Unmetabolized Folic Acid; Pediatrics
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: This research project will consist of a clinical trial in which children with SCD are randomly selected to initially receive 1 mg per day of folic acid (the current standard dose) or a placebo for a 12-week period. Following that, each participant will have a 12 week wash-out period and then treatments are reversed (folic acid supplement or placebo) for 12 weeks. No controls are included in the study as each participant serves as their own control during periods of no supplementation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind clinical trials, so neither participants nor medical care providers will be aware of the participants group assignment in order to limit bias, changes in dietary habits, or medical treatment. The outcomes assessor will also be unaware of participant assignment in order to limit bias in analysis of samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folic Acid Supplement [Phase 1] (Other): Phase 1: Folic acid supplement (1 mg per day) for 12 weeks; Phase 2: Wash-out period (no supplement or placebo) for 12 weeks; Phase 3: Placebo for 12 weeks
  Interventions: Dietary Supplement: Folic Acid Supplement; Dietary Supplement: Placebo
- Placebo [Phase 1] (Other): Phase 1: Placebo for 12 weeks; Phase 2: Wash-out period (no supplement or placebo) for 12 weeks; Phase 3: Folic acid supplement (1 mg per day) for 12 weeks
  Interventions: Dietary Supplement: Folic Acid Supplement; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Folic Acid Supplement — 1 milligram folic acid
Dietary Supplement: Placebo — Placebo

SUMMARY:
Folic acid supplementation (1mg/d) is the standard recommendation for Canadian children with Sickle cell disease (SCD), even though it can provide up to six times the recommended intake amount for healthy children. There is growing concern that too much folic acid can be detrimental to health as high folate levels and circulating unmetabolized folic acid (UMFA), which occurs in blood with doses of folic acid as low as 0.2mg/d, have been associated with accelerated growth of some pre-cancerous cells, and altered DNA methylation and gene expression.

To inform the efficacy and potential harm of high-dose folic acid supplementation in Canadian children with SCD, a double-blind randomized controlled cross-over trial is proposed. Children with SCD (n=36, aged 2-19 y) will be recruited from BC Children's Hospital and randomized to initially receive 1 mg/d folic acid or a placebo for 12-weeks (wk). After a 12-wk washout period, treatments will be reversed.

DETAILED DESCRIPTION:
Blood samples will be collected at baseline and 12-wk of each treatment period (weeks 12, 24, and 36).

Serum and RBC concentrations of total folate, different folate forms and clinical outcomes will be measured at baseline and after each treatment period. Dietary folate intake will be assessed at baseline.

The objective of this study is to determine efficacy and potential harm of folic acid supplementation, versus no supplementation, in Canadian children with sickle cell disease.

It is hypothesized that: (1) there will be no difference in mean RBC folate concentrations across folic acid and placebo groups after 12-wk, (2) none of the participants will have folate deficiency, and (3) compared to periods of no supplementation, during periods of high-dose folic acid supplementation participants will show no difference in clinical outcomes, but have higher plasma unmetabolized folic acid concentrations.

Significance: There is a need to determine if the current clinical practice of high-dose folic acid supplementation is efficacious, and warranted.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with SCD aged 2-19 y attending British Columbia Children's Hospital
* Individuals having received routine daily supplementation of folic acid for the prior 12-weeks

Exclusion Criteria:

* Individuals receiving a blood transfusion in the prior 12-weeks
* Individuals allergic to any components of the supplement (cellulose, methylcellulose, magnesium stearate, and/or titanium dioxide)
* Individuals presenting with megaloblastic anemia in the prior 12-weeks
* Individuals with pulmonary, renal and/or cardiac complications (severe or recurrent acute chest syndrome)
* Individuals routinely taking medications known to interfere with B vitamin metabolism (chloramphenicol, methotrexate, metformin, sulfasalazine, phenobarbital, primidone, triamterene, barbiturates)
* Individuals who are currently pregnant, planning to become pregnant in the next 9-months, or currently breastfeeding
* Individuals who have participated in a clinical research trial in the previous 30 days
* Individuals who have donated blood in the previous 30 days
* Individuals with unstable medical conditions or unstable laboratory results.

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Red Blood Cell Folate Concentration | 12 weeks
  Biochemical folate status marker (nmol/L)
Red Blood Cell Folate Concentration | 36 weeks
  Biochemical folate status marker (nmol/L)

SECONDARY OUTCOMES:
Serum Folate Concentration | 12 weeks
  Biochemical folate status marker (nmol/L)
Serum Folate Concentration | 36 weeks
  Biochemical folate status marker (nmol/L)
Plasma Unmetabolized Folic Acid Concentration | 12 weeks
  Biochemical folate marker (nmol/L)
Plasma Unmetabolized Folic Acid Concentration | 36 weeks
  Biochemical folate marker (nmol/L)
S-adenosyl-methionine Concentration | 12 weeks
  Biochemical folate metabolite (µmol/L)
S-adenosyl-methionine Concentration | 36 weeks
  Biochemical folate metabolite (µmol/L)
S-adenosyl-homocysteine Concentration | 12 weeks
  Biochemical folate metabolite (µmol/L)
S-adenosyl-homocysteine Concentration | 36 weeks
  Biochemical folate metabolite (µmol/L)
Total homocysteine Concentration | 12 weeks
  Biochemical folate metabolite (µmol/L)
Total homocysteine Concentration | 36 weeks
  Biochemical folate metabolite (µmol/L)
Acute Pain Crises | 12 weeks
  Participant self-reported occurrence (# of episodes, and severity of episodes)
Acute Pain Crises | 36 weeks
  Participant self-reported occurrence (# of episodes, and severity of episodes)
Megaloblastic anemia | 12 weeks
  Determined by hemoglobin and Mean Corpuscular Volume (MCV) concentrations below/above age-specific hematological cut-offs
Megaloblastic anemia | 36 weeks
  Determined by hemoglobin and Mean Corpuscular Volume (MCV) concentrations below/above age-specific hematological cut-offs

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Karakochuk, PhD, RD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published articles, after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Access will be available starting within 3 months of the publication of results and up to a period of 5 years
Access Criteria: Researchers who provide a methodologically sound proposal may gain access following receipt of a signed data access agreement.

REFERENCES:
- [Background] Williams BA, McCartney H, Adams E, Devlin AM, Singer J, Vercauteren S, Wu JK, Karakochuk CD. Folic acid supplementation in children with sickle cell disease: study protocol for a double-blind randomized cross-over trial. Trials. 2020 Jun 29;21(1):593. doi: 10.1186/s13063-020-04540-7. PMID 32600389
- [Derived] Williams BA, McCartney H, Singer J, Devlin AM, Vercauteren S, Amid A, Wu JK, Karakochuk CD. Folic acid supplementation in children with sickle cell disease: a randomized double-blind noninferiority cross-over trial. Am J Clin Nutr. 2025 Apr;121(4):910-920. doi: 10.1016/j.ajcnut.2025.02.001. Epub 2025 Feb 5. PMID 39921095
- See also: Study protocol — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-020-04540-7